CLINICAL TRIAL: NCT05813496
Title: A Multicenter, Interventional, Two-arm, Parallel-group, Randomized, Double-blinded, Placebo-controlled, Phase IV Trial to Evaluate the Efficacy of Alpha-Lipoic Acid in the Treatment of Symptomatic Diabetic Polyneuropathy in Egypt
Brief Title: Phase IV Trial to Evaluate Efficacy of Alpha-Lipoic Acid in Treating Symptomatic Diabetic Polyneuropathy in Egypt
Acronym: MIRACLE-ALA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eva Pharma (Industry)
Collaborators: MARC-CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Cl_Tr_17122019
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Polyneuropathy, Diabetic
Keywords: Thiotacid; Double-blinded; Placebo-controlled; Multi-center
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid; Tablets

STUDY DESIGN:
Intervention Model Description: After signing the ICF, eligible patients were randomized in a 1:1 allocation ratio, into one of the two treatment groups, to receive either ALA or placebo. Randomization will be done using an interactive web response system (IWRS).
  Randomization was stratified by baseline body mass index (BMI) (< 25 Kg/m2 or 25-40 Kg/m2) followed by age (<45 years or ≥ 45 years) and gender (male or female).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IND Arm (Experimental): 200 patients will receive one tablet of 600 mg of alpha-lipoic acid twice a day orally for 24 weeks.
  Interventions: Drug: Alpha-Lipoic Acid (ALA)
- Placebo Arm (Placebo Comparator): 200 patients will receive one tablet of placebo twice a day orally for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alpha-Lipoic Acid (ALA) — Oral tablet
  Other Names: Thiotacid® 600 mg
  Arms: IND Arm
Drug: Placebo — Microcrystalline cellulose (Ph 101) 427.5 mg, Magnesium stearate 71.25 mg, Sodium laurayl sulphate 6 mg, Croscarmellose sodium 11.25 mg, Silica, colloid anhydrous 11.25 mg, and Purified talc 30 mg.
  Other Names: Oral tablet
  Arms: Placebo Arm

SUMMARY:
The purpose of the study is to find out whether ALA is effective and safe for treating Egyptian diabetic patients with symptomatic polyneuropathy. The ADA stated that despite the exploration of several pharmacological therapies for DPN management, substantial evidence on medicines that modify the natural history of DPN is still absent. This is a multicenter, interventional, two-arm, parallel-group, randomized, double-blinded, placebo-controlled, phase IV trial. Patients will be administered either one tablet of placebo or one tablet containing 600 mg of ALA twice a day for 24 weeks, depending on the randomization process.

DETAILED DESCRIPTION:
This is a multicenter, interventional, two-arm, parallel-group, randomized, double-blinded, placebo-controlled, phase IV trial to evaluate the efficacy and safety of ALA in the treatment of diabetic patients with symptomatic polyneuropathy in Egypt.

Patients will be randomly assigned to receive either :

* One tablet of 600 mg ALA twice a day orally for 24 weeks. Total daily dose during the study duration (24 weeks) = 1200 mg. , or
* One tablet of placebo twice a day orally for 24 weeks.
* The standard of Care (SOC) treatments will be prescribed for both study arms (Experimental and control arm) as per the routine clinical practice and following the relevant clinical guidelines. The SOC treatments include those for glycemic control and other treatments for the management of painful diabetic polyneuropathy; when needed through the course of the clinical study. As per the ADA and NICE guidelines (ADA, 2022) ("Type 2 Diabetes Adults Manag.," 2022); Pregabalin, Duloxetine, or Gabapentin are recommended as initial pharmacologic treatments for neuropathic pain in diabetes.

Estimated recruitment period: 24 weeks Estimated duration of participation: 24 weeks of treatment in addition to a screening period of approximately 1 week Visit 1: Screening/Baseline visit Visit 2: After 4 weeks ± 5 days of treatment Visit 3 (Phone call 1): After 12 weeks ± 15 days of treatment Visit 4 (Phone call 2): After 20 weeks ± 15 days of treatment Visit 5: After 24 weeks ± 15 days of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Male or female patients aged ≥ 18 and ≤ 64 years.
3. Type 2 diabetes mellitus (T2DM) patients as defined according to the American Diabetes Association (ADA) criteria with diabetes duration ≥ 1 year.
4. Hemoglobin A1c (HbA1c) ≤10%.
5. Patients with symptomatic distal symmetrical polyneuropathy (DSPN) attributable to diabetes; after a thorough evaluation for other causes of neuropathy, with evidence of polyneuropathy based on abnormal peripheral nerve function according to clinical and electrophysiological examinations.
6. Patients treated with oral antidiabetic drugs and/or insulin.
7. Patients with the treatment regimen, weight, diet, and physical activity level relatively acceptable as judged by the investigator within 1 month prior to study entry.
8. Patients with working telephone numbers.

Exclusion Criteria:

1. Female patients with child-bearing potential not using effective birth control methods including oral contraceptives with a stable regimen for at least 2 months, depo-medroxyprogesterone, a barrier method alone (diaphragm, condoms, or contraceptive sponge with spermicidals), or an intrauterine device that has been in place for at least 2 months.
2. Patients with neuropathies other than DSPN; myopathy and other neurologic diseases that might interfere with the assessment of the severity of DSPN.
3. Patients with a recent history of drug or alcohol abuse; within 1 year prior to study entry.
4. Patients with a history of peripheral vascular disease and/or foot ulcers.
5. Patients with a history of organ transplantation.
6. Patients with a history of cardiovascular, pulmonary, gastrointestinal, hematologic, or endocrine disease, or malignancy that cause neuropathic pain.
7. Hospitalization due to hypoglycemia or ketoacidosis within 3 months prior to study entry.
8. Patients with significant hepatic or renal disease [Serum creatinine > 1.8 mg/dL for men and > 1.6 mg/dL for women, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 times upper limit of normal (ULN)].
9. Use of medications indicated for neuropathic pain relief within 15 days (washout period) prior to study entry. For analgesia, standard doses of salicylates, ibuprofen, indoles, fenamates, oxicams, or pyrazoles are allowed.
10. Use of antioxidants (including but not limited to vitamin E, vitamin C, and β-carotene) or pentoxifylline within 1 month prior to study entry.
11. Use of medications or vitamins known to cause peripheral neuropathy including but not limited to the use of phenytoin or carbamazepine over 15 or more years, or use of pyridoxine > 100 mg/d within 12 months prior to study entry.
12. Use of ≥ 50 mg ALA or use of alpha-linolenic acid-containing substances within 3 months prior to study entry.
13. Use of an investigational drug within 6 months prior to study entry.
14. Enrollment in any other clinical trial during the time of this trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
To compare the relative change in NCS parameters between the study arms | After four weeks of treatment
  The main objective of this study is to calculate the efficacy of alpha-lipoic acid in comparison with placebo in diabetic patients with symptomatic polyneuropathy assessed by the change in NCS parameters after 4 weeks of treatment using student t-test (Mann-Whitney test for non-parametric data) to compare relative change between treatment arm and control arm. This analysis will be comparative and will be done on eligible subjects without protocol violation and who have at least one treatment dose and an evaluable primary endpoint.

SECONDARY OUTCOMES:
To compare the relative change in NCS parameters between the study arms. | After 24 weeks of treatment
  The efficacy of alpha-lipoic acid in comparison with placebo in diabetic patients with symptomatic polyneuropathy assessed by the change in NCS after 24 weeks of treatment using student t-test (Mann-Whitney test for non-parametric data) to compare relative change between treatment arm and control arm.
To compare the relative change in NDS and Neuro-QoL between the study arms. | After 24 weeks of treatment
  The efficacy of alpha-lipoic acid in comparison with placebo in diabetic patients with symptomatic polyneuropathy as assessed by the change in NDS* total score (out of 10 = the sum of the scores for right and left sides) using student t-test (Mann-Whitney test for non-parametric data) to compare relative change between treatment and control arms.
To compare the frequency of the need to rescue analgesic medications between the study arms | After 24 weeks of treatment
  The efficacy alpha-lipoic acid in comparison with placebo in diabetic patients with symptomatic polyneuropathy assessed by number of patients receiving rescue analgesic medications using chi square test to compare between treatment arm and control arm. This analysis will be comparative and will be done on eligible subjects without protocol violation and who have at least one treatment dose and evaluable primary endpoint
To assess safety of Thiotacid® as per the nature and severity of the recorded adverse events. | After 24 weeks of treatment
  The safety of alpha-lipoic acid in diabetic patients with symptomatic neuropathy assessed by the number of patients experiencing AE/SAE and number of patients who discontinued study drug due to AEs. These will be described using counts/percentages with 95% CI. This analysis will be descriptive and will be conducted on all patients enrolled to the study who signed an ICF.

CONTACTS AND LOCATIONS:
Overall Officials: Samir H Assaad Khali, PhD, Principal Investigator — Alexandria University Hospital / Internal Medicine; Mohamed R Halawa, PhD, Principal Investigator — Ain-Shams University Hospital / Internal Medicine; Nabil AF El Kafrawy, PhD, Principal Investigator — Menoufia University Hospital / Internal Medicine; Hanan M El Sotouhy Gawish, PhD, Principal Investigator — Mansoura University Hospital / Internal Medicine; Khaled ES El Hadidy, PhD, Principal Investigator — Beni Suef University Hospital / Internal Medicine
Locations (5):
- Egypt (5):
  - Alexandria University, Alexandria, Bab Sharqi
  - Beni Suef University Hospital, Banī Suwayf, Beni Suweif Governorate
  - Ain-Shams University Hospital, Cairo, Heliopolis
  - Menoufia University Hospital, Shibīn al Kawm, Shebin El Kom
  - Mansoura University Hospital, Al Mansurah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ADA. (2022). Standards of Medical Care in Diabetes-2022 Th E Jou R Nal of C Li N Ical an D Appli Ed R Esearc H an D Education. Diabetes Care, 45(Suppliment 1), S1-S264. https://doi.org/10.2337/dc22-SREV
- [Background] Boulton AJ, Vinik AI, Arezzo JC, Bril V, Feldman EL, Freeman R, Malik RA, Maser RE, Sosenko JM, Ziegler D; American Diabetes Association. Diabetic neuropathies: a statement by the American Diabetes Association. Diabetes Care. 2005 Apr;28(4):956-62. doi: 10.2337/diacare.28.4.956. No abstract available. PMID 15793206
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Roman-Pintos LM, Villegas-Rivera G, Rodriguez-Carrizalez AD, Miranda-Diaz AG, Cardona-Munoz EG. Diabetic Polyneuropathy in Type 2 Diabetes Mellitus: Inflammation, Oxidative Stress, and Mitochondrial Function. J Diabetes Res. 2016;2016:3425617. doi: 10.1155/2016/3425617. Epub 2016 Dec 12. PMID 28058263
- [Background] Type 2 diabetes in adults: management. (2022). Type 2 Diabetes in Adults: Management, March. https://www.ncbi.nlm.nih.gov/books/NBK553486/
- [Background] Young MJ, Boulton AJ, MacLeod AF, Williams DR, Sonksen PH. A multicentre study of the prevalence of diabetic peripheral neuropathy in the United Kingdom hospital clinic population. Diabetologia. 1993 Feb;36(2):150-4. doi: 10.1007/BF00400697. PMID 8458529
- [Background] Ziegler D, Gries FA. Alpha-lipoic acid in the treatment of diabetic peripheral and cardiac autonomic neuropathy. Diabetes. 1997 Sep;46 Suppl 2:S62-6. doi: 10.2337/diab.46.2.s62. PMID 9285502